CLINICAL TRIAL: NCT01661946
Title: Systemic Absorption of Bevacizumab and Ranibizumab in Humans Treated for Diabetic Macular Edema
Brief Title: Bloodstream Absorption of Avastin and Lucentis After Injection Into the Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Sanjay Sharma, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QueensU
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Macular Edema
Keywords: vascular endothelial growth factor; macular edema; diabetic retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Active Comparator): intravitreal injection of 0.5mg ranibizumab in usual fashion
  Interventions: Drug: Ranibizumab
- Bevacizumab (Active Comparator): intravitreal injection of 1.25mg bevacizumab in usual fashion
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is an off-label but cheaper treatment for diabetic macular edema.
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Ranibizumab — Ranibizumab is a vascular endothelial growth factor inhibitor designed for ocular use
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
Currently, two similar medications are available for injection into the eye to treat a variety of eye diseases. These medications are called ranibizumab (Lucentis) and bevacizumab (Avastin). They both have a similar mechanism of action and work equally well, however only ranibizumab was designed for use in the eye. It is significantly more expensive per injection than bevacizumab (by a factor of roughly 40x).

In published studies trends have been noted towards an increased rate of systemic side effects such as heart attacks and strokes. This is presumably due to absorption of the drug(s) from the eye into the bloodstream, however this has never been shown before. The purpose of the investigators study was to compare the bloodstream levels of bevacizumab and ranibizumab at various time points after injection into the eye. This required the creation of a sophisticated assay to measure blood levels of the drugs.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* patients in whom anti-vascular endothelial growth factor (VEGF) therapy is indicated for the treatment of diabetic macular edema
* able to return for extra clinic visits according to study schedule

Exclusion Criteria:

* active malignancy
* previous retinal laser treatment
* previous anti-VEGF therapy
* previous vitrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sharma, MD MBA MSc FRCSC, Principal Investigator — Department of Ophthalmology, Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab | Bevacizumab
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Ranibizumab | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 62.5 [50 to 73] | 67.9 [55 to 85] | 65.2 [50 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Anti-VEGF Antibody
Description: The serum concentrations of anti-VEGF antibody (bevacizumab or ranibizumab) will be measured pre-injection as well as at various time points after injection (1 day, 1 week, 2 weeks, 1 month). These time points are selected based on previously completed animal studies. The Cmax will be compared between bevacizumab and ranibizumab.
Time Frame: 1 month
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ranibizumab | Bevacizumab
Number analyzed (Participants) | 5 | 5
ng/mL | 25.22 (7.59) | 9.56 (2.50)

ADVERSE EVENTS:
Arm/Group | Ranibizumab | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No